CLINICAL TRIAL: NCT05073276
Title: Non-Weight Bearing Versus Partial Controlled Weightbearing During the First Six Weeks of Rehabilitation After Multiple Knee Ligament Reconstruction: a Randomized Controlled Trial
Brief Title: Non- Vs Partial Controlled Weightbearing After Multiple Knee Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Twin Cities Orthopedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RFL_NWB vs PWB-Multi-Knee Lig
Record Dates: First submitted 2021-09-13; First posted 2021-10-11 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Knee Injuries
Keywords: anterior cruciate ligament (ACL); Multiple Knee Ligament Reconstruction
MeSH Terms: conditions — Knee Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-weightbearing for the first six weeks after surgery (Active Comparator): Not weightbearing after surgery
  Interventions: Other: Physical Therapy
- Partial weight -bearing for the first six weeks after surgery (Experimental): Partial weightbearing will be defined as 40% of the patient's body weight.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Patient is randomized to the weightbearing group the day after surgery.

SUMMARY:
This is a prospective randomized controlled trial with the purpose to determine if patients undergoing isolated posterior cruciate ligament (PCL) reconstruction, or isolated medial collateral ligament (MCL) reconstruction, or combined PCL, anterior cruciate ligament (ACL), fibular collateral ligament (FCL), posterolateral corner (PLC), and MCL reconstructions (or any combination of multiple ligaments) can safely begin partial controlled weightbearing for the first six weeks after surgery.

DETAILED DESCRIPTION:
Patients will be randomly assigned to one of two rehabilitation protocols for the first six weeks post-surgery:

1. non-weightbearing
2. partial weightbearing

An immobilizer brace in extension will be used from post-operative day 0 through 4 and a dynamic stabilizing posterior knee brace (Ossur) will be used from 5 days through 6 months post-surgery to protect against increased posterior translation forces due to gravity and while weightbearing for patients with PCL reconstructions.

Specific Aims

1. Primary Aim: To determine if there is clinical equivalence in millimeters of posterior tibial translation on posterior stress radiographs at six months post-surgery between patients who are non-weightbearing versus partial controlled weightbearing during the first six weeks of post-surgical rehabilitation.
2. Primary Aim: To determine if there is clinical equivalence in millimeters of valgus and/or varus compartment gapping on stress radiographs at six months post-surgery between patients who are non-weightbearing versus partial controlled weightbearing during the first six weeks of post-surgical rehabilitation.
3. Secondary Aim: To determine if there is a difference in pain, edema, range of motion, gait, and quadriceps strength between groups.

The current standard of care for posterior cruciate ligament reconstruction and multiligament reconstruction is non-weightbearing for the first six weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 14 years old, <60
* Reconstruction of PCL alone
* Reconstruction of MCL alone
* Reconstruction of combined multiligament injuries (PCL+ (FCL, PLC, ACL, MCL))
* Reconstruction of multiligament injuries (ACL+MCL)
* Males or females
* Is willing and able to comply with the clinical trial plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

* < 14 years old
* >60 years old
* Pregnant
* Revision PCL reconstructions
* Previous or concurrent vascular injury (vascular bypass procedure)
* Associated fractures requiring concurrent surgery
* Concurrent meniscal root or radial repair surgery

Ages: 14 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Gapping (mm) measured on Standard of Care Varus stress radiographs | Pre-operative
  stress radiographs
Gapping (mm) measured on Standard of Care Varus stress radiographs | 6 months post-surgery
  stress radiographs

SECONDARY OUTCOMES:
Numeric Pain Scale (NPS) (0-10 rating) | Baseline and 6 months
  Pain scale 0-100
Measurements by physical therapists (Edema, thigh circumference) | 4,7, and 10 months after surgery
  Measurements with tape
Measurements by physical therapists (range of motion) | 4,7, and 10 months after surgery
  Measurements with goniometer
Measurements by physical therapists (Quadriceps strength, gait analysis) | 4,7, and 10 months after surgery
  Measurements by biomechanics lab
Patient reported outcome scores | Baseline, 3 months, 6 months, 1 year
  Surveys: International Knee Documentation Committee (IKDC), Cincinnati Knee Rating System (Cincinnati), Knee injury and Osteoarthritis Outcome Score (KOOS), Tegner, Lysholm Knee Scoring Scale (Lysholm), and Veterans Rand 12 (VR-12) or Short Form-12 (SF-12) General Health Survey, lower extremity functional scale, Sports Medicine Questionnaire and survey/patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Robert F LaPrade, MD, PhD, Principal Investigator — Twin Cities Orthopedics
Locations (1):
- Twin Cities Orthopedics, Edina, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No